CLINICAL TRIAL: NCT00387504
Title: Phase I Trial of Intravenous Fenretinide (4-HPR) for Patients With Malignant Solid Tumors
Brief Title: Fenretinide in Treating Patients With Metastatic or Unresectable Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: California Cancer Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000508770; U01CA062505 (NIH); CCC-PHI-54; NCI-7540
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Fenretinide

INTERVENTIONS:
Drug: fenretinide — 4-HPR (Fenretinide) is given as a continuous intravenous infusion (CIV) for five consecutive days. Cycle is repeated every 3 weeks, if PR, CR or stable disease for 6 cycles.
Other: pharmacological study — samples drawn per protocol

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fenretinide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of fenretinide in treating patients with metastatic or unresectable malignant solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of fenretinide in patients with metastatic or unresectable malignant solid tumors.
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics and in vivo activity of this drug in these patients.
* Determine, preliminarily, disease or tumor response in patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive fenretinide IV continuously on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete or partial response may continue to receive fenretinide at the discretion of the study chair.

Cohorts of 3-6 patients receive escalating doses of fenretinide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Patients undergo blood sample collection to determine plasma concentrations (pharmacokinetics) of fenretinide periodically during course 1 and at the end of courses 2-6.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 21 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor malignancy

  * Metastatic and/or unresectable disease
* No standard curative or palliative measures exist or remain effective
* Measurable or evaluable disease
* No known brain metastases unless previously resected or irradiated with no treatment with steroids for more than 1 month

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy > 3 months
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (5 times ULN for patients with known liver metastases)
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for ≥ 6 months after completion of study treatment
* No uncontrolled diabetes mellitus at high risk for hypertriglyceridemia (i.e., fasting serum glucose concentration > 200 mg/dL OR hemoglobin A1C > 7.5%)
* No egg allergy
* No history of allergic reactions to compounds of similar chemical or biologic composition to fenretinide (e.g., isotretinoin, vitamin A, or tretinoin)
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude compliance with study requirements
* No known hypertriglyceridemia requiring medication
* No identified familial hyperlipidemia disorder

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* Prior treatment with oral fenretinide is allowed provided no severe toxicity occurred
* At least 2 weeks since prior major surgery
* More than 4 weeks since prior chemotherapy or radiotherapy

  * At least 6 weeks since prior nitrosoureas or mitomycin C
* No other concurrent investigational agents
* No other concurrent anticancer chemotherapy
* No other concurrent antioxidants*
* No concurrent hormone-ablative agents, including steroids, except for adrenal replacement or anti-inflammatory indications
* No other concurrent anticancer agents or therapies
* No concurrent herbal or other alternative therapies*
* No concurrent vitamin supplements (e.g., vitamin A, ascorbic acid, or vitamin E)*

  * Standard-dose multivitamin allowed
* No other concurrent medications that may act as modulators of intracellular ceramide levels or ceramide cytotoxicity, sphingolipid transport, p-glycoprotein, multidrug resistance protein 1 (MRP1), or MRP1 drug/lipid transporters, including any of the following*:

  * Cyclosporine or any of its analogues
  * Verapamil
  * Tamoxifen or its analogue
  * Ketoconazole
  * Chlorpromazine
  * Mifepristone
  * Indomethacin
  * Sulfinpyrazone NOTE: *Patients who have discontinued these drugs for ≥ 1 week are eligible
* No concurrent medications that may cause pseudotumor cerebri, including any of the following:

  * Tetracycline
  * Nalidixic acid
  * Nitrofurantoin
  * Phenytoin
  * Sulfonamides
  * Lithium
  * Amiodarone
* No concurrent total parenteral nutrition (TPN) with intralipids
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2006-11; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of fenretinide | at end of study
Toxicity as measured by type (organ affected or laboratory determination such as absolute neutrophil count), severity (NCI CTCAE v3.0), time of onset (course number), duration, and reversibility or outcome | ongoing
Survival and time to failure as measured by Kaplan-Meier | at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, MD, Study Chair — University of Southern California
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - City of Hope Medical Group, Pasadena, California
  - University of California Davis Cancer Center, Sacramento, California
  - Texas Tech University Health Sciences Center, Lubbock, Texas